CLINICAL TRIAL: NCT00721578
Title: An Observational Study Of Patients Receiving Therapy For Systemic Fungal Infections
Brief Title: A Study Of Indian Patients Receiving Therapy For Systemic Fungal Infections
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A1501089
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Systemic Fungal Infections
Keywords: Observational study; Effectiveness; Safety; Tolerability; Systemic Fungal Infection
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — Patients must have received (in the Intensive Care Unit [ICU] at study entry) at least 1 day therapy with systemic antifungal agent for treatment of a proven or suspected fungal infection. The decision regarding choice of antifungal agent would lie with the treating physician and will necessarily precede and be independent of the decision to enroll a patient into the study.
  Other Names: Vfend

SUMMARY:
To collect and summarize information on the diagnosis, management, and clinical and mycological outcomes of patients with systemic fungal infections in order to better understand the effectiveness of antifungals in the treatment of Systemic Fungal Infections (SFI) in India.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for enrollment in the study database, patients must have received (in the Intensive Care Unit [ICU] at study entry) at least 1 day therapy with systemic antifungal agent for treatment of a proven or suspected fungal infection.

Exclusion Criteria:

* None.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A database of outcomes in patients with proven or probable Systemic Fungal Infections (SFI) treated with antifungals in 5 centers across India.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- India (2):
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, New Delhi, New Delhi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501089&StudyName=An%20Observational%20Study%20Of%20Patients%20Receiving%20Therapy%20For%20Systemic%20Fungal%20Infections

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole Antifungal Treatment; Other Antifungal Treatment: Systemic antifungals were administered based on approved prescribing documents and were adjusted solely according to medical and therapeutic necessity. The choice of systemic antifungal agent was dependent on the investigators decision and was independent of enrollment into the study.
Period: Overall Study
Arm/Group | Voriconazole Antifungal Treatment | Other Antifungal Treatment
Started | 12 | 11
Completed | 10 | 9
Not Completed | 2 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Systemic antifungals were administered based on approved prescribing documents and were adjusted solely according to medical and therapeutic necessity. The choice of systemic antifungal agent was dependent on the investigators decision and was independent of enrollment into the study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis of Systemic Fungal Infection (SFI)
Description: Evidence of clinical signs and symptoms of systemic fungal infection including: fever, hypotension, or radiological or microbiological evidence, as assessed by the investigator.
Time Frame: Up to 9 months
Population: Full analysis set (FAS) = all enrolled participants who received at least one dose of antifungal therapy. n = number of participants who had microbiological assessments performed. SOT = start of treatment, EOT = end of treatment
Measure: Number; unit: Participants
Groups:
- All Antifungal Therapies: Systemic antifungals were administered based on approved prescribing documents and were adjusted solely according to medical and therapeutic necessity. The choice of systemic antifungal agent was dependent on the investigators decision and was independent of enrollment into the study
Arm/Group | All Antifungal Therapies
Number analyzed (Participants) | 23
Participants
  Fever | 20
  Hypotension | 6
  Radiological Assessment (SOT - Abnormal) | 18
  Radiological Assessment (EOT - Abnormal) | 3
  Microbiological Assessment (positive, n=7) | 5
  Microbiological Assessment (negative, n=7) | 2

2. Primary Outcome: Management of SFI: Choice of Treatment
Description: Number of participants treated with each antifungal therapy. Each participant may have recieved 1 or more treatments as deemed clinically necessary by the investigator.
Time Frame: Up to 9 months
Population: FAS.
Measure: Number; unit: Participants
Arm/Group | All Antifungal Therapies
Number analyzed (Participants) | 23
Participants
  Voriconazole | 12
  Fluconazole | 11
  Caspofungin acetate | 3
  Amphotericine B, liposome | 3
  Amphotericin B | 2
  Caspofungin | 1

3. Primary Outcome: Management of SFI: Reason for Selection of Antifungal Agent
Description: Number of participants with reason for investigator's selection of particular antifungal therapy.
Time Frame: Up to 9 months
Population: FAS. Data were not analyzed.
Measure: Number; unit: Participants
Groups:
- Therapy for Systemic Fungal Infections: Systemic antifungals were administered based on approved prescribing documents and were adjusted solely according to medical and therapeutic necessity. The choice of systemic antifungal agent was dependent on the investigators decision and was independent of enrollment into the study
Arm/Group | Therapy for Systemic Fungal Infections
Number analyzed (Participants) | 0

4. Primary Outcome: Total Daily Dose for Selected Antifungal Agent
Time Frame: Up to 9 months
Population: FAS. Data were not analyzed.
Measure: Number; unit: mg
Arm/Group | Therapy for Systemic Fungal Infections
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With Clinical Outcomes.
Description: Clinical outcomes, as assessed by the investigator, defined as:
  Cured: clinical signs and symptoms of fungal infection absent. Improved: clinical signs and symptoms of fungal infection improved. Stable: no change in overall clinical findings, compared with previous reporting period.
  Deteriorated: clinical signs and symptoms of fungal infection worsened (including death).
  Indeterminate; clinical signs and symptoms of fungal infection were insufficient to make an evaluation.
Time Frame: Up to 9 months
Population: FAS.
Measure: Number; unit: Participants
Arm/Group | Therapy for Systemic Fungal Infections
Number analyzed (Participants) | 23
Participants
  Cured | 2
  Improved | 11
  Stable | 6
  Deteriorated | 4

6. Primary Outcome: Number of Participants With Mycological Outcomes
Description: Mycological outcome of persistence (continued presence of fungi on microbiology despite therapy), eradication (absence of fungi after therapy
  ), or unknown (results are not available/not known) as assessed by the Investigator/Physician.
Time Frame: Up to 9 months
Population: FAS.
Measure: Number; unit: Participants
Arm/Group | Therapy for Systemic Fungal Infections
Number analyzed (Participants) | 23
Participants
  Persistence | 3
  Eradication | 8
  Unknown | 11
  Not Recorded | 1

7. Secondary Outcome: Concomitant Medications
Time Frame: Up to 9 months
Population: FAS.
Measure: Number; unit: Participants
Arm/Group | Therapy for Systemic Fungal Infections
Number analyzed (Participants) | 23
Participants
  Acetorphan | 1
  Acetylcysteine | 3
  Acetylsalycilic acid | 2
  Acetylsalicylic acid/clopidogrel | 1
  Aciclovir | 1
  Allopurinol | 1
  Ambroxol | 1
  Ambroxol Hydrochloride | 1
  Amikacin | 4
  Amiodarone Hydrochloride | 2
  Amlodipine | 1
  Atorvastatin | 1
  Atracurium | 1
  B-Komplex "Leciva" | 1
  Breva | 1
  Budesonide | 2
  Carvedilol | 1
  Cefazolin | 1
  Cefepime | 1
  Cefotaxime | 1
  Cefotaxime/sulbactam | 1
  Ciprofloxacin | 1
  Clindamycin | 2
  Clopidogrel | 2
  Colistin mesilate sodium | 2
  Cordalin/old form/ | 2
  Deflazacort | 1
  Diltiazem hydrochloride | 1
  Doripenem | 1
  Doxofylline | 1
  Enalapril maleate | 1
  Enoxaparin | 1
  Epoetin alfa | 1
  Escitalopram | 1
  Esomeprazole | 2
  Esomeprazole magnesium | 1
  Ethambutol | 2
  Fludrocortisone | 1
  Fluoxetine hydrochloride | 1
  Folic acid | 1
  Folinic acid | 1
  Furosemide | 2
  Granulocyte colony stimulating factor | 1
  Haloperidol | 2
  Heparin-fraction, sodium salt | 6
  Hydrocortisone | 1
  Hydrocortisone hydrogen succinate | 4
  Imipenem | 2
  Immunoglobulins | 1
  Insulin glargine | 1
  Isoniazid | 1
  Lactulose | 2
  Lekovit ca | 2
  Levetiracetam | 2
  Levocetirizine | 1
  Levofloxacin | 4
  Linezolid | 4
  Meropenem | 8
  Methylprednisolone | 2
  Metoclopramide hydrochloride | 3
  Metronidazole | 5
  Moxifloxacin | 1
  Mycophenolate mofetil | 1
  Ofloxacin | 1
  Ondansetron | 4
  Pantoprazole | 9
  Pantoprazole sodium | 6
  Paracetamol | 8
  Pazufloxacin | 1
  Pheniramine maleate | 1
  Phenobarbital | 1
  Phenytoin sodium | 2
  Pip/tazo | 1
  Piperacillin | 1
  Piperacillin/tazobactam | 4
  Polybion | 2
  Polymyxin B | 2
  Polymyxin B sulfate | 3
  Potassium | 2
  Prednisolone | 2
  Primaxin | 1
  Propylthiouracil | 1
  Prulifloxacin | 1
  Pyridoxine | 1
  Ramipril | 2
  Ranolazine | 1
  Ribolac | 1
  Sertraline | 2
  Simvastatin | 1
  Solifenacin | 1
  Sulperazon | 5
  Teicoplanin | 11
  Tienam | 1
  Tramadol | 3
  Valproic acid | 1
  Vancomycin | 1
  Vancomycin hydrochloride | 1
  Vitamin B-complex | 1
  Vitamin B12 (cyanocobalamin and derivatives) | 1

8. Secondary Outcome: Median Duration of Antifungal Therapy
Time Frame: Up to 9 months
Population: FAS.
Measure: Median (Full Range); unit: Days
Groups:
- Therapy for Systemic Fungal Infection: Systemic antifungals were administered based on approved prescribing documents and were adjusted solely according to medical and therapeutic necessity. The choice of systemic antifungal agent was dependent on the investigators decision and was independent of enrollment into the study
Arm/Group | Therapy for Systemic Fungal Infection
Number analyzed (Participants) | 23
Days
  All Antifungals | 12.0 [4 to 127]
  Voriconazole | 13.0 [5 to 127]

9. Secondary Outcome: Medication Administration
Description: Participants who received medication by IV or oral administration, reported by total number of participants receiving IV and total number of participants receiving oral administation (overall), and by total number of participants receiving voriconazole only by IV or oral administration.
Time Frame: Up to 9 months
Population: FAS.
Measure: Number; unit: Participants
Arm/Group | Therapy for Systemic Fungal Infections
Number analyzed (Participants) | 23
Participants
  All Antifungals Intravenous | 17
  All Antifungals Oral | 11
  Voriconazole Intravenous | 5
  Voriconazole Oral | 6

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Therapy for Systemic Fungal Infections
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 3/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapy for Systemic Fungal Infections (N=23)
Pancreatitis (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 3
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Coma (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapy for Systemic Fungal Infections (N=23)
Vomiting (Gastrointestinal disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Primary and Secondary outcome measured were arbitrarily defined as they were not defined in the protocol.

This study was terminated prematurely due to slow recruitment rate leading to a small (23) number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.